CLINICAL TRIAL: NCT06682533
Title: Efficacy and Tolerability of 14-Day Tegoprazan-based Triple Therapy for Eradication of Helicobacter Pylori Eradication: A Retrospective Study
Brief Title: Tegoprazan- Versus PPI-based H. Pylori Eradication
Status: Recruiting | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2024-11
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: H.Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PPI-BID group: Standard dose of PPI bid, amoxicillin 1000 mg bid, clarithromycin 500 mg bid, tripotassium dicitrate bismuthate (DENOL) 300 mg bid 14 days
- Tegoprazan-BID group: Tegoprazan 50 mg bid, amoxicillin 1000 mg bid, clarithromycin 500 mg bid, tripotassium dicitrate bismuthate (DENOL) 300 mg bid for 14 days
- PPI-QID group: Standard dose of PPI bid, amoxicillin 500 mg qid, clarithromycin 500 mg bid, tripotassium dicitrate bismuthate (DENOL) 300 mg bid 14 days
- Tegoprazan-QID group: Tegoprazan 50 mg bid, amoxicillin 500 mg qid, clarithromycin 500 mg bid,tripotassium dicitrate bismuthate (DENOL) 300 mg bid for 14 days

SUMMARY:
In 2015, vonoprazan, a potassium-competitive blocker (P-CAB), was launched in Japan and used as an alternative for proton pump inhibitors (PPIs) for eradicating Helicobacter pylori. In recent studies, vonoprazan-based triple therapy significantly increased the eradication rate from 72.8% to 87.9%, compared to PPI treatment group. Accordingly, the Japanese Helicobacter treatment guidelines recommend prescribing P-CAB for eradication treatment. In 2018, a new P-CAB, tegoprazan, was developed in Korea and approved for gastric ulcer treatment. Subsequently, it was proven effective in the treatment of reflux esophagitis compared to PPIs in a non-inferiority clinical trial. P-CAB can increase the gastric pH to 6 or higher within 7 hours after taking tegoprazan. Because tegoprazan can be taken after meals, it can improve patient compliance for H. pylori eradication. Unlike vonoprazan in Japan, however, tegoprazan-based eradication in Korean population was similar to conventional PPI-based treatment. To date, the eradication success rates of PPI and tegoprazan-based triple therapy were 76.4-84.2% and 77.3-84.3%, respectively, and there was no significant difference between the two treatment groups.

Bismuth has long been used as a semi-metal in the dyspepsia and traveler's diarrhea. In H. pylori eradication therapy, several guidelines recommended the addition of bismuth to treatment regimens. Recently, bismuth was added to the 2-week triple regimen to increase the first-line H. pylori eradication rate in countries with high antibiotic resistance. The H. pylori eradication significantly increased from 87.5-88.1% to 95.8-97.3% in a recent study. The odds ratio was 1.63-2.18 in bismuth-added treatment group, compared to no use of bismuth group. In subgroup analysis, odd ratio was 1.66-2.22 in high clarithromycin-resistant areas. However, there was no comparative analysis of PPIs and tegoprazan in a bismuth-added triple therapy.

DETAILED DESCRIPTION:
The investigators aim to evaluate the eradication success rate and treatment compliance between PPI and tegoprazan in first-line H. pylori treatment with adding bismuth.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* Drug allergy to antibiotics
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rates | 6 weeks
  Urea breath test after completing H. pylori eradication regimen

SECONDARY OUTCOMES:
Treatment compliance | 6 weeks
  Assessment of patients' numbers completing H. pylori eradication regimen
Drug-related adverse event rate | 6 weeks
  Bitter tongue, nausea/vomiting, bloating, diarrhea, and abdominal pain during H. pylori treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No